CLINICAL TRIAL: NCT02812329
Title: Intervention to Encourage HIV Testing and Counseling Among Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Digitalmill (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1604017531
Record Dates: First submitted 2016-06-21; First posted 2016-06-24 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

ARMS (1):
- HIV prevention videogame (Experimental): Participants will play PlayForward on a tablet computer for 1 hour, two times per week for 3 weeks.
  Interventions: Behavioral: HIV prevention videogame

INTERVENTIONS:
Behavioral: HIV prevention videogame — Assess acceptability and efficacy of a HIV prevention videogame

SUMMARY:
This study aims to minimize risk of human immunodeficiency virus (HIV) in adolescent boys and girls, ages 15-16, by promoting HIV testing and counseling (HTC) through the use of an interactive videogame. With input from focus groups of adolescents, the investigators will adapt an HIV prevention videogame, PlayForward: Elm City Stories, for adolescents ages 15-16 . The investigators will then pilot test the videogame in 30 adolescents to assess the acceptability and feasibility of the videogame. They will also assess whether the videogame increased the participants' intentions to obtain HTC, whether they actually obtained HTC, and whether the videogame increased knowledge of HIV.

DETAILED DESCRIPTION:
Adolescents are at high risk of contracting human immunodeficiency virus (HIV). To help them to minimize their risk and maintain their uninfected status, it is critical to give them the information, motivation, and skills to get HIV testing and counseling (HTC).

The current proposal focuses on adapting an existing HIV prevention videogame, PlayForward: Elm City Stories (R01HD062080), developed for 11-14 year olds, to include a primary focus on promoting access to and uptake of HTC in adolescent boys and girls, ages 15-16. PlayForward, an engaging and interactive videogame grounded in social learning theory and the theory of planned behavior, was developed through extensive work with its target audience to focus on the delay of sexual initiation in young teens and is currently demonstrating preliminary efficacy in a large randomized controlled trial (RCT).

In this Phase I proposal, PlayForward will be adapted for use in a slightly older age group with the primary outcome of encouraging them (increasing intentions) to obtain HTC and increasing knowledge about HIV/AIDS.

Working with the multi-disciplinary team of the play2PREVENT (p2P) Lab, we will conduct the formative work with our target audience and content experts to modify PlayForward for a focus on promoting HTC. To this end, our specific aims for this Phase I proposal targeting HTC in 15-16 year old adolescents are to:

Aim 1: Translate our culturally and socially-tailored videogame PlayForward to focus on HTC in an older age group of 15-16 year old boys and girls by:

1. Developing a conceptual model of the theoretical mechanisms of behavior change to be applied specifically within the game. We will develop this model with input from 4 focus groups of 5 adolescents each (n = 20, aged 15-16) and the extant literature.
2. This model will inform the development of a set of intervention manuals ("Game Playbooks") targeting the new outcome.

   Aim 2: Modify aspects of the PlayForward game to reflect this new focus by pilot testing it with 30 adolescents, aged 15-16 to determine in a pre-post design:
3. The intervention's acceptability and feasibility using self-report data on the game play experience.
4. Preliminary evidence of the efficacy of the intervention by collecting data on i) intentions to seek HTC; ii) actual obtaining of HTC; and iii) knowledge about HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* participants must: 1) be 15-16 years of age and 2) be able to participate in a mobile videogame (willing to sit with a tablet computer for 60 minutes/session to play the game).

Exclusion Criteria:

-

Ages: 15 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of a HIV prevention videogame measured by self-report questionnaire developed by the study team, | After 3 weeks of using the videogame
  Efficacy measure will include items on intentions around HIV Testing/Counseling and knowledge of HIV.
Efficacy of a HIV prevention videogame measured by self-report questionnaire developed by the study team. | Three weeks after 3 weeks of using the videogame
  Efficacy measure will include items on intentions around HIV Testing/Counseling and knowledge of HIV.

SECONDARY OUTCOMES:
Satisfaction/acceptability of the HIV prevention videogame measured by self-report questionnaire developed by the study team. | After 3 weeks of using the videogame

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E. Fiellin, M.D., Principal Investigator — Yale University